CLINICAL TRIAL: NCT00788203
Title: The Development of an Early Intervention for the Prevention of Childhood Obesity
Brief Title: Prevention of Childhood Obesity
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: W. Stewart Agras, MD. Principal Investigator, Stanford University
Other Study IDs: SU-11052008-1335; R21HD055637 (NIH)
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 5-keys program: Counseling re family feeding behaviors.
- Lifestyle counseling: Counseling re healthy eating for child and family

SUMMARY:
This study is conducting preliminary testing to find out whether a particular educational program can alter parental overcontrol of their children's eating. There is evidence from previous studies that children who are irritable, cry a lot, tend to be overcontrolled and are at high risk for developing overweight. If the education program can change parental behavior the next study would examine whether this affects children's weight over a longer period of time.

DETAILED DESCRIPTION:
There are two main studies in this project. For both studies families with a child between 2 and 4-years will be entered to the study although only the parents will participate. At least one parent will be overweight with a BMI>27.5, and the child will have a reactive temperament assessed by the Children's Behavior Questionnaire (CBQ) completed by the parent with a combined score on the approach/impulsivity scales of 4.65 (possible range 1 - 7). The cut-points for parental BMI and their child's temperament derive from our previous prospective risk factor study. Screening will consist of a brief telephone screen to ascertain willingness to participate in further screening and self-reported BMI. Both parents will be invited to the laboratory to ascertain whether they meet BMI criteria. In Study 1 parents with a child with either reactive or non-reactive temperament patterns will be entered to this study. In Study 2 only parents with a child with a reactive temperament will be admitted to the study. There will be no randomization in Study 1. There will also be 2 focus groups each lasting 90-minutes to ascertain typical child feeding problems, and a pilot administration of the interventions. In Study 2 parents will be randomized to receive either the experimental intervention or a health education program aimed at enhancing their children's health. Each group session will last 90-minutes and there will be 10 group sessions at weekly intervals. Assessments in both studies will be similar and will consist of questionnaires aimed at assessing family and children's feeding behaviors and parental attitudes and behaviors concerning their own weight/shape and dieting. We estimate that the assessments will take approximately 60-minutes to complete in Study 1 and 45-minutes each in Study 2 because extraneous questions will be removed as a result of findings in Study 1.

ELIGIBILITY:
Inclusion Criteria:

For study 1, 60 families (120 parents) with a child between the age of 2-4 years will be entered to the study. Children of these families will be at risk for overweight because the family will contain at least one obese parent. For study 2, 100 families (200 parents) will be entered to the study. Children of these families will be at risk for overweight and have a reactive temperament. The reason for using this population is that a combination of parental obesity and a child with a reactive temperament appears to put the child at high risk for the development of overweight.

Exclusion Criteria:Parental exclusions:

1. Not able to comprehend English well enough to participate in assessments or the intervention.
2. Serious non-obesity related physical illness, (e.g., cancer), which would preclude participation in assessment or intervention.
3. Serious current psychiatric disorder, e.g. schizophrenia, uncontrolled bipolar disorder, mental retardation that would preclude participation in assessment or intervention.
4. Single parents

Child exclusions:

1. Serious physical illness or related treatments that would affect feeding or weight including history of feeding aversion, failure to thrive, and use of nasogastric or gastrostomy feeding.
2. Prematurity below 37-weeks associated with prolonged hospitalization, ongoing need for nutritional supplementation, or naso-gastric feeding.(parental report)
3. Serious current developmental problems including any that might interfere with self-feeding or require additional parental feeding support e.g. developmental delay, autism. (parental report).

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 2-4 years at risk for overweight with at least one overweight/obese parent
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Parental restraint concerning eating | Prospective

SECONDARY OUTCOMES:
Daily eating pattern | Weekly
  Parental report of feeding frequency

CONTACTS AND LOCATIONS:
Overall Officials: William Stewart Agras, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States